CLINICAL TRIAL: NCT02119559
Title: Assessment of Circulating Tumor Cells as an Early Predictive Marker of Response to a First Line Treatment Based on an Anti-Human Epidermal Growth Factor Receptor (HER), Cetuximab, in Patients With Inoperable Recurrent and/or Metastatic Head-and-neck Squamous-cell Carcinoma.
Brief Title: Circulating Tumor Cells as an Early Predictive head-and -Neck Squamous-cell Carcinoma
Acronym: CIRCUTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 8825; ID-RCB:2011-A01174-37 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2014-03-28; First posted 2014-04-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2012-09

CONDITIONS: Metastatic Head-and-neck Squamous-cell Carcinoma
Keywords: Circulating Tumor Cells; Treatment Efficiency; Biomarker
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTC assay, Cetuximab (Other): Detection & characterization of viable CTC in the peripheral blood.
  Interventions: Other: Blood analysis by EPISPOT and CellSearch®

INTERVENTIONS:
Other: Blood analysis by EPISPOT and CellSearch®
  Other Names: A counting of CTC using three technologies: EPISPOT, CellSearch®, flow cytometer sorter/analyzer.

SUMMARY:
In France, the incidence of head and neck squamous cell carcinomas (HNSCC) is 16 000 new cases/year. During these last years, many new chemotherapies and targeted therapies have been developed improving significantly the overall survival of patients notably anti-HER molecules. In inoperable recurrent and/or metastatic HNSCC, the best treatment is based on an anti-Human Epidermal Growth Factor Receptor (EGFR) antibody, targeting Human Epidermal Growth Factor Receptor 1 (HER1), the Cetuximab combined with platinum +/- 5 Fluoro Uracil (5FU): " Extreme protocol ". However, no clinical or biological criteria predictive of drug efficacy have been reported yet. Thus, the development of such a predictive factor is an urgent need in HNSCC at both the clinical and pharmacy-economic level, to propose the best personalized treatment. One idea would be to enumerate and characterize the circulating tumor cells (CTC) which could give us an early evaluation of the therapeutic efficiency. In this context, the investigators have developed an innovative technology, the EPISPOT assay (patent of the University Medical Center of Montpellier), that allows the detection & characterization of viable CTC in the peripheral blood. The EPISPOT technology has been already evaluated in the breast and prostate cancer.Thus, the investigators would like for the first time to perform a prospective study on a cohort of patients treated following the Extreme protocol, with this technology, to assess the predictive value of CTC count. The investigators will use the CellSearch® system as the reference test.

DETAILED DESCRIPTION:
This is a multi-centric prospective non randomized open labeled study performed on a cohort of patients with inoperable recurrent and/or metastatic HNSCC who will be treated, with a first line treatment based on an anti-Human Epidermal Growth Factor Receptor (HER), the Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yo.
* Histologically or cytologically confirmed recurrent and/or metastatic Squamous Cell Carcinoma Head and Neck (SCCHN) (excluding nasopharyngeal carcinoma) not suitable for local therapy : surgery and/or radiotherapy ; or metastatic disease with or without primary evolving tumor.
* Target definable with Response Evaluation Tumors Criteria in Solid (RECIST) 1.1 criteria.
* WHO performance status 0,1 or 2.
* Life expectancy > 3 month at inclusion.
* Patient eligible for first line chemotherapy based on cisplatin (100 mg/m2 as a 1-hour intravenous (IV) infusion on day 1) or carboplatin (AUC 5 mg/ml.min by 1-hour IV infusion, day 1) and an infusion of 5-FU (1000 mg/m2/day for 4 days) every 3 weeks, with cetuximab (initial dose of 400 mg/m2 [2-hour IV infusion] followed by subsequent weekly doses of 250 mg/m2 [1-hour IV infusion], ending at least 1 hour before the start of chemotherapy).
* Consent form for participation signed.

Exclusion Criteria:

* Other chemotherapy protocol not involving platinum and cetuximab.
* Other proven synchronous evolving cancer.
* Evolving infectious disease or severe other disease preventing the patient from receiving treatment.
* Patient refusal.
* Patient unable to consent.
* Pregnant or breastfeeding, or premenopausal women not taking effective contraception.
* Current Participation to other clinical trial except experimental molecules.
* Vulnerable persons protected by law.
* People under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Predictive value of the CTC on the Progression Free Survival | Duration study 2 years
  The primary outcome aims to evaluate the predictive value of the early progression of the CTC performed with the EPISPOT assay on the progression free survival in a cohort of patients treated with protocol "Extreme". The progression disease is assessed based on imagery techniques.

SECONDARY OUTCOMES:
Prognostic value of the CTC at baseline (EPISPOT) and to compare for the first time the results with those obtained with the CellSearch system. | Duration study 2 years
Prognostic value of the CTC at baseline (EPISPOT) | Duration study 2 years
Predictive value of the early progression of CTC (EPISPOT) on the overall survival | Duration study 2 years
Compare for the first time the results with those obtained with the CellSearch® system | Duration study 2 years
Evaluate the expression of EGFR in CTCs before and after administration of cetuximab (Erbitux) with both technologies and EPISPOT CellSearch ® | Duration study 2 years
Evaluate the impact of the presence of epithelial-mesenchymal transition (EMT) marker on the prognosis | Duration study 2 years

CONTACTS AND LOCATIONS:
Overall Officials: RENAUD GARREL, MD, Principal Investigator — CHU GUI DE CHAULIAC
Locations (1):
- Department of Otorhinolaryngology, CHU Gui de Chauliac, Montpellier, France

REFERENCES:
- [Derived] Garrel R, Mazel M, Perriard F, Vinches M, Cayrefourcq L, Guigay J, Digue L, Aubry K, Alfonsi M, Delord JP, Lallemant B, Even C, Daures JP, Landais P, Cupissol D, Alix-Panabieres C. Circulating Tumor Cells as a Prognostic Factor in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma: The CIRCUTEC Prospective Study. Clin Chem. 2019 Oct;65(10):1267-1275. doi: 10.1373/clinchem.2019.305904. Epub 2019 Aug 6. PMID 31387885
- [Derived] Le Louedec F, Alix-Panabieres C, Lafont T, Allal BC, Garrel R, Digue L, Guigay J, Cupissol D, Delord JP, Lallemant B, Alfonsi M, Aubry K, Mazel M, Becher F, Perriard F, Chatelut E, Thomas F. Cetuximab pharmacokinetic/pharmacodynamics relationships in advanced head and neck carcinoma patients. Br J Clin Pharmacol. 2019 Jun;85(6):1357-1366. doi: 10.1111/bcp.13907. Epub 2019 Apr 13. PMID 30811063